CLINICAL TRIAL: NCT02818764
Title: Pathophysiology of Delirium in Patients Undergoing Total Hip Arthroplasty: Role of Intraoperative Cerebral Perfusion and EEG Abnormalities
Brief Title: Delirium, Intraoperative Cerebral Perfusion and EEG Abnormalities After Total Hip Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: COVID related limitations
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 822008
Record Dates: First submitted 2016-06-02; First posted 2016-06-30 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Delirium; Hip Arthroplasty; Elderly
Keywords: serum biomarkers; cerebral blood flow; modified Blessed Dementia Rating scale; Confusion Assessment Method; Delirium Rating Scale-98
MeSH Terms: conditions — Delirium | interventions — Blood Specimen Collection; Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Cerebral Spinal Fluid (CSF)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Delirium: Subjects undergoing elective total joint arthroplasty determined to have delirium by post operative 3D-CAM.
  Data collected on intraoperative cerebral blood flow and oxygen extraction fraction.
  CSF collected for biomarkers. Blood colelcted for biomarkers.
  Interventions: Procedure: Blood Draw; Procedure: Cerebral Spinal Fluid collection; Device: Electroencephalogram; Device: Cerebral blood flow and oxygen extraction fraction
- Non-delirium: Subjects undergoing elective total joint arthroplasty determined not to have delirium by post oeprative 3D-CAM.
  Data collected on intraoperative cerebral blood flow and oxygen extraction fraction.
  CSF collected for biomarkers. Blood colelcted for biomarkers.
  Interventions: Procedure: Blood Draw; Procedure: Cerebral Spinal Fluid collection; Device: Electroencephalogram; Device: Cerebral blood flow and oxygen extraction fraction

INTERVENTIONS:
Procedure: Blood Draw — 5 mL of blood from the patients preoperative, postoperative, 1 day and 2 days after surgery for a total of 20 mL.
Procedure: Cerebral Spinal Fluid collection — Fluid collected at the time of dural puncture if patients will undergo spinal anesthesia
  Other Names: CSF
Device: Electroencephalogram — Test used to detect abnormalities related to electrical activity of the brain will be done during surgery.
  Other Names: EEG
Device: Cerebral blood flow and oxygen extraction fraction — NIRS measurement of Cerebral blood flow and cerebral tissue oxygen concentration.

SUMMARY:
The overall objective of this study is to test for perturbations in intraoperative electroencephalogram (EEG) , cerebral blood flow (CBF), cerebral metabolic rate of oxygen consumption (CMRO2), oxygen extraction fraction (OEF), and serum and cerebral spinal fluid biomarkers associated with delirium in high risk population having elective hip arthroplasty at Penn Presbyterian Medical Center (PPMC).

DETAILED DESCRIPTION:
All prospective patients will be given a copy of the informed consent which explains the details and responsibilities of the study.

Each patient will have a preoperative baseline 3D-CAM and MOCA to document preoperative cognitive function and possible criteria for exclusion.

1. The 3D -Confusion Assessment Method (CAM) test is a clinician evaluation and algorithm for the binary determination of presence or absence of delirium.
2. Montreal Confusion Assessment (MOCA) - to be given preoperatively to determine if element of pre-existing cognitive impairment

Intraoperatively each patient will have a NIR Optode patch placed to measure intraoperative cerebral blood flow and oxygen extraction fraction and cerebral metabolic rate of oxygen consumption.

A non-invasive frontal EEG patch will be placed prior to or at the start of anesthesia. Anesthetic depth will be measured using the SEDline® by Masimo. Continuous raw EEG, spectral edge, compressed spectral analysis and percentage suppressed will be recorded from the SEDline® monitor.

The investigators will be drawing blood from patients who agree to participate in the study. Preoperative blood sampling will be done while the investigators place the intravenous line, or if present, from an arterial line.

If a spinal anesthetic is being used, 5 mL of cerebral spinal fluid (CSF) will be collected at the time of dural puncture prior to the administration of the neuraxial blockade.

Members of the research team will administer 3D-CAM testing on post-operative days 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 65 years of age and over scheduled for elective total joint arthroplasty
2. Mentally competent and able to give consent for enrollment in the study
3. Patients at any age with a pre-existing diagnosis of dementia or acquired cognitive deficit. Consented by legally authorized representative (LAR).

Exclusion Criteria:

1. Patients currently delirious
2. Acute neurological disease like stroke or brain tumor
3. Current alcohol or substance abuse at risk of postoperative withdrawal

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing total joint arthroplasty who are 65 years of age and older.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-06; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Delirium Rating Scale | change from Baseline through day 2 post op
  The severity of delirium in this patient population as quantified by the DRS
Serum biomarkers | change from Baseline through day 2 post op
  The change in serum biomarkers S100β in patients who are diagnosed with delirium by DRS.

SECONDARY OUTCOMES:
Change in cerebral blood flow | change from Baseline through 3 hours
  Changes in CBF from the norm in the patients who develop delirium
Confusion Assessment Method | change from Baseline through day 2 post op
  Changes in patient performance to determine the presence or absence of delirium as measured by the CAM test

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Kofke, MD MBA FCCM, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Trzepacz PT, Mittal D, Torres R, Kanary K, Norton J, Jimerson N. Validation of the Delirium Rating Scale-revised-98: comparison with the delirium rating scale and the cognitive test for delirium. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):229-42. doi: 10.1176/jnp.13.2.229. PMID 11449030
- [Background] Fong TG, Bogardus ST Jr, Daftary A, Auerbach E, Blumenfeld H, Modur S, Leo-Summers L, Seibyl J, Inouye SK. Cerebral perfusion changes in older delirious patients using 99mTc HMPAO SPECT. J Gerontol A Biol Sci Med Sci. 2006 Dec;61(12):1294-9. doi: 10.1093/gerona/61.12.1294. PMID 17234823
- [Background] Gokgoz L, Gunaydin S, Sinci V, Unlu M, Boratav C, Babacan A, Soncul H, Halit V, Inanir S, Ersoz A. Psychiatric complications of cardiac surgery postoperative delirium syndrome. Scand Cardiovasc J. 1997;31(4):217-22. doi: 10.3109/14017439709041749. PMID 9291540
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Blessed G, Tomlinson BE, Roth M. The association between quantitative measures of dementia and of senile change in the cerebral grey matter of elderly subjects. Br J Psychiatry. 1968 Jul;114(512):797-811. doi: 10.1192/bjp.114.512.797. No abstract available. PMID 5662937